CLINICAL TRIAL: NCT00279318
Title: Consortium for Identification of Environmental Triggers of Type 1 Diabetes
Brief Title: TEDDY - The Environmental Determinants of Diabetes in the Young
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH); Juvenile Diabetes Research Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DK095300; DK100238; DK106955; 1UC4DK095300-01 (NIH); 1UC4DK100238-01 (NIH); 1UC4DK106955-01 (NIH); 1UC4DK112243-01 (NIH); 1UC4DK117483-01 (NIH); 1U01DK124166-01 (NIH); 1U01DK128847-01 (NIH)
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Environment; Exposures; Diet; Toxins; Psychosocial; Infectious Agents; Bacterial; Viral; Immunizations; Autoantibody
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, PBMCs, stool, urine, saliva, nasal swabs, nail clippings, water, teeth
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Population, First Degree Relative: Newborns with high risk HLA in the general population or having a first-degree relative affected with T1DM.

SUMMARY:
The long-term goal of the TEDDY study is the identification of infectious agents, dietary factors, or other environmental agents, including psychosocial factors which trigger T1DM in genetically susceptible individuals or which protect against the disease. Identification of such factors will lead to a better understanding of disease pathogenesis and result in new strategies to prevent, delay or reverse T1DM.

DETAILED DESCRIPTION:
Epidemiologic patterns suggest that viruses, nutrition, toxic agents or socioeconomic psychosocial factors may contribute to the etiology alone or in combination. Elucidation is confounded by the long interval between exposure and onset of clinical disease, as well as the interaction of multiple genes and/or insults, which appear to interact in a complex manner. Numerous studies have investigated environmental influences but have yielded conflicting results. This may be in part due to the failure to account for genetic susceptibility, begin observation at early ages or in utero, and/or monitor subjects long term and frequently.

Hypotheses:

1. Initiation of persistent beta-cell autoimmunity and progression from beta-cell autoimmunity to diabetes is increased with:

   1. Exposure to a trigger factor during pregnancy, such as infections, preeclampsia, blood incompatibility, or birth weight.
   2. Differences in the timing of the introduction and/or the type of dietary constituents that include exposure to cereals or gluten, exposure to cow's milk during infancy and/or childhood, and short duration of breast- feeding;
   3. Lower intake of serum 25 hydroxyvitamin D in early infancy, vitamin E, anti-oxidants (e.g., carotenoids, ascorbic acid, selenium, or omega-3 fatty acids);
   4. Higher frequency of specific (e.g., enterovirus, rotavirus, or bacterial) infections, or non-specific childhood infections including those that exhibit molecular mimicry;
   5. Increased exposure to routine childhood immunizations and their timing;
   6. Environmental factors that may be contained in drinking water (e.g., low concentrations of zinc or high concentrations of nitrates, or lower pH levels);
   7. Exposure to household pets, and various allergies;
   8. Excessive weight gain;
   9. Increased psychological stress.
2. The risk of persistent beta-cell autoimmunity is lower in children from the general population than in offspring or siblings of T1DM patients when stratifying for the HLA DR-DQ genotype and exposure to environmental triggers.
3. The interaction of HLA DR-DQ genotype with exposure to dietary or infectious factors leads to increased incidence of beta-cell autoimmunity and T1DM.
4. We expect that in some families study participation will be associated with affective (anxiety, depression) and behavioral responses (e.g. actions to prevent possible T1DM).

ELIGIBILITY:
Inclusion Criteria:

* Newborns with high risk HLA in the general population or having a first- degree relative affected with T1DM
* Newborns are less than 4 months of age

Exclusion Criteria:

* Have an illness or birth defect that precludes long-term follow-up or involves use of treatment that may alter the natural history of diabetes (e.g. steroids or insulin)
* Refuses to have blood and stool samples stored at the NIDDK Repository

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Childen up to 4 months of age with specified HLA are enrolled and followed longitudnally until 15 years of age
Sampling Method: Non-Probability Sample
Enrollment: 8667 (Actual)
Dates: Start 2004-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Appearance of one or more islet cell autoantibodies: GADA, IAA, or IA-2A confirmed at two consecutive visits. | September 2025

SECONDARY OUTCOMES:
Development of T1DM | September 2025

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P. Krischer, PhD, Principal Investigator — University of South Florida; Marian J. Rewers, MD, PhD, Principal Investigator — University of Colorado Health Science Center; William A. Hagopian, MD, PhD, Principal Investigator — Pacific Northwest Research Institute; Ake Lernmark, MD, PhD, Principal Investigator — Lund University; Jorma Toppari, MD, PhD, Principal Investigator — Wellbeing Services County of Southwest Finland; Richard McIndoe, PhD, Principal Investigator — Augusta University Research Institute, Inc.; Anette G. Ziegler, MD, Principal Investigator — Diabetes Research Institute; Beena Akolkar, PhD, Study Director — National Institutes of Diabetes and Digestive Kidney Diseases
Locations (7):
- United States (4):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Augusta University, Gainesville, Florida
  - Augusta University, Augusta, Georgia
  - Pacific Northwest Research Institute, Seattle, Washington
- Wellbeing Services County of Southwest Finland, Turku, Finland
- Diabetes Research Institute, Munich, Germany
- Lund University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository https://repository.niddk.nih.gov/studies/teddy/?query=teddy
URL: https://repository.niddk.nih.gov/studies/teddy/?query=teddy

REFERENCES:
- [Derived] Kyronniemi A, Valtanen T, Koskenniemi J, Vahasalo P, Harkonen T, Ilonen J, Toppari J, Knip M, Veijola R. Extremely Early Appearance of Islet Autoantibodies in Genetically Susceptible Children. Pediatr Diabetes. 2023 Dec 11;2023:9973135. doi: 10.1155/2023/9973135. eCollection 2023. PMID 40303239
- [Derived] Gesualdo P, Melin J, Karban R, Crouch C, Killian M, Hopkins D, Adamsson A, Stock J, Johnson SB, Baxter J; TEDDY Study Group. Structures and strategies for retaining an international pediatric cohort from birth: Lessons from The Environmental Determinants of Diabetes in the Young (TEDDY) study. Contemp Clin Trials Commun. 2025 Jan 23;44:101405. doi: 10.1016/j.conctc.2024.101405. eCollection 2025 Apr. PMID 40027280
- [Derived] Euren A, Lynch K, Lindfors K, Parikh H, Koletzko S, Liu E, Akolkar B, Hagopian W, Krischer J, Rewers M, Toppari J, Ziegler A, Agardh D, Kurppa K; TEDDY Study Group. Risk of celiac disease autoimmunity is modified by interactions between CD247 and environmental exposures. Sci Rep. 2024 Oct 26;14(1):25463. doi: 10.1038/s41598-024-75496-w. PMID 39462122
- [Derived] Gesualdo P, Melin J, Karban R, Crouch C, Killian M, Hopkins D, Adamsson A, Stock J, Johnson SB, Baxter J. Structures and Strategies for Retaining an International Pediatric Cohort from Birth: Lessons from The Environmental Determinants of Diabetes in the Young (TEDDY) Study. Res Sq [Preprint]. 2024 Jun 6:rs.3.rs-4421364. doi: 10.21203/rs.3.rs-4421364/v1. PMID 38883796
- [Derived] Melin J, Lynch KF, Lundgren M, Aronsson CA, Larsson HE, Johnson SB. Factors assessed in the first year of a longitudinal study predict subsequent study visit compliance: the TEDDY study. Eur J Med Res. 2023 Dec 15;28(1):592. doi: 10.1186/s40001-023-01563-z. PMID 38102669
- [Derived] Krischer JP, Liu X, Lernmark A, Hagopian WA, Rewers MJ, She JX, Toppari J, Ziegler AG, Akolkar B; TEDDY Study Group. Predictors of the Initiation of Islet Autoimmunity and Progression to Multiple Autoantibodies and Clinical Diabetes: The TEDDY Study. Diabetes Care. 2022 Oct 1;45(10):2271-2281. doi: 10.2337/dc21-2612. PMID 36150053
- [Derived] Melin J, Lynch KF, Lundgren M, Aronsson CA, Larsson HE, Johnson SB; TEDDY Study Group. Is staff consistency important to parents' satisfaction in a longitudinal study of children at risk for type 1 diabetes: the TEDDY study. BMC Endocr Disord. 2022 Jan 10;22(1):19. doi: 10.1186/s12902-021-00929-w. PMID 35012530
- [Derived] Krischer JP, Liu X, Lernmark A, Hagopian WA, Rewers MJ, She JX, Toppari J, Ziegler AG, Akolkar B; TEDDY Study Group. Characteristics of children diagnosed with type 1 diabetes before vs after 6 years of age in the TEDDY cohort study. Diabetologia. 2021 Oct;64(10):2247-2257. doi: 10.1007/s00125-021-05514-3. Epub 2021 Jul 22. PMID 34291312
- [Derived] Johnson RK, Tamura R, Frank N, Uusitalo U, Yang J, Niinisto S, Andren Aronsson C, Ziegler AG, Hagopian W, Rewers M, Toppari J, Akolkar B, Krischer J, Virtanen SM, Norris JM; TEDDY Study Group. Maternal food consumption during late pregnancy and offspring risk of islet autoimmunity and type 1 diabetes. Diabetologia. 2021 Jul;64(7):1604-1612. doi: 10.1007/s00125-021-05446-y. Epub 2021 Mar 30. PMID 33783586
- [Derived] Frank NM, Lynch KF, Uusitalo U, Yang J, Lonnrot M, Virtanen SM, Hyoty H, Norris JM; TEDDY Study Group. The relationship between breastfeeding and reported respiratory and gastrointestinal infection rates in young children. BMC Pediatr. 2019 Sep 18;19(1):339. doi: 10.1186/s12887-019-1693-2. PMID 31533753
- [Derived] Hippich M, Beyerlein A, Hagopian WA, Krischer JP, Vehik K, Knoop J, Winker C, Toppari J, Lernmark A, Rewers MJ, Steck AK, She JX, Akolkar B, Robertson CC, Onengut-Gumuscu S, Rich SS, Bonifacio E, Ziegler AG; TEDDY Study Group; Teddy Study Group. Genetic Contribution to the Divergence in Type 1 Diabetes Risk Between Children From the General Population and Children From Affected Families. Diabetes. 2019 Apr;68(4):847-857. doi: 10.2337/db18-0882. Epub 2019 Jan 17. PMID 30655385
- [Derived] Hagopian WA, Erlich H, Lernmark A, Rewers M, Ziegler AG, Simell O, Akolkar B, Vogt R Jr, Blair A, Ilonen J, Krischer J, She J; TEDDY Study Group. The Environmental Determinants of Diabetes in the Young (TEDDY): genetic criteria and international diabetes risk screening of 421 000 infants. Pediatr Diabetes. 2011 Dec;12(8):733-43. doi: 10.1111/j.1399-5448.2011.00774.x. Epub 2011 May 12. PMID 21564455
- See also: TEDDY Study Public site — http://teddy.epi.usf.edu/